CLINICAL TRIAL: NCT06716151
Title: A Phase I, Randomized, Double-blind, Placebo-controlled, Single/mulit Dose-escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of HB0034 in Adult Healthy Subjects
Brief Title: A Study to Evaluate HB0034 in Healthy Chinese Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Huaota Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HB0034-HV-01-03
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Healthy subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Active Comparator: HB0034 dose group 1 (Experimental): 6 subjects receive a single-dose of HB0034, a recombinant humanized anti-IL-36R IgG1 monoclonal antibody
  Interventions: Drug: HB0034
- Active Comparator: HB0034 dose group 2 (Experimental): 6 subjects receive a single-dose of HB0034, a recombinant humanized anti-IL-36R IgG1 monoclonal antibody
  Interventions: Drug: HB0034
- Active Comparator: HB0034 dose group 3 (Experimental): 6 subjects receive a single-dose of HB0034, a recombinant humanized anti-IL-36R IgG1 monoclonal antibody
  Interventions: Drug: HB0034
- Active Comparator: HB0034 dose group 4 (Experimental): 6 subjects receive a single-dose of HB0034, a recombinant humanized anti-IL-36R IgG1 monoclonal antibody
  Interventions: Drug: HB0034
- Active Comparator: HB0034 dose group 5 (Experimental): 6 subjects receive a single-dose of HB0034, a recombinant humanized anti-IL-36R IgG1 monoclonal antibody
  Interventions: Drug: HB0034
- Active Comparator: HB0034 dose group 6 (Experimental): 8 subjects receive a multi-dose of HB0034, a recombinant humanized anti-IL-36R IgG1 monoclonal antibody
  Interventions: Drug: HB0034
- Active Comparator: HB0034 dose group 7 (Experimental): 8 subjects receive a multi-dose of HB0034 a recombinant humanized anti-IL-36R IgG1 monoclonal antibody
  Interventions: Drug: HB0034
- Placebo group (Placebo Comparator): 17 subjects receive placebo
  Interventions: Drug: HB0034 matching placebo

INTERVENTIONS:
Drug: HB0034 — Recombinant Humanized Anti-IL-36R Monoclonal antibody
  Arms: Active Comparator: HB0034 dose group 1; Active Comparator: HB0034 dose group 2; Active Comparator: HB0034 dose group 3; Active Comparator: HB0034 dose group 4; Active Comparator: HB0034 dose group 5; Active Comparator: HB0034 dose group 6; Active Comparator: HB0034 dose group 7
Drug: HB0034 matching placebo — HB0034 matching Palcebo
  Arms: Placebo group

SUMMARY:
The aim of this study is to investigate the safety and tolerability of HB0034 in healthy subjects following a single dose or multiple dose.

DETAILED DESCRIPTION:
This study consisted of a single-dose escalation study and a multi-dose escalation study to evaluate the safety, tolerability, pharmacokinetics, and immunogenicity of HB0034 in Chinese healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects age ≥ 18 and ≤ 55 years.
* Body Mass Index (BMI) ≥ 17.5 and ≤ 32 kg/m².
* Normal ECG, blood pressure, respiratory rate, temperature, and heart rate, unless the investigator considers any abnormality to be not clinically significant.

Signed and dated written informed consent prior to admission to the study in accordance with GCP and local legislation.

Exclusion Criteria:

- History of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, psychiatric, or neurological disease.

Current or history of malignancy. • Family history of premature Coronary Heart Disease (CHD)

* History of clinically significant opportunistic infection (e.g., invasive candidiasis or pneumocystis pneumonia).
* Pregnant or Breasting feeding subject. Women with a positive pregnancy test.
* Further exclusion criterias apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with drug related adverse events (AEs) | up to 113 days
  An AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the investigational drug

SECONDARY OUTCOMES:
Cmax | Up to 113 days
  The maximum measured concentration of the analysis in plasma
AUC0-infinity | up to 113 days
  The area under the concentration-time curve of the analysis in plasma over the time interval from 0 extrapolated to infinity

CONTACTS AND LOCATIONS:
Locations (1):
- Central Hospital affiliated to Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided